CLINICAL TRIAL: NCT04970056
Title: Pancreatic Cancer Early Detection Consortium
Acronym: PRECEDE
Status: Recruiting | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Responsible Party: Sponsor
Other Study IDs: PRECEDE
Record Dates: First submitted 2021-04-21; First posted 2021-07-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-06

CONDITIONS: Pancreas Cancer; Pancreas Cyst; Pancreatic Ductal Adenocarcinoma; Genetic Predisposition
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A standardized procedure for collection and processing of human blood will be applied to all blood samples collected as part of the study. Barcoded samples will be stored at the clinical centers, and corresponding data will be entered into the study database. Any protocol deviations should also be recorded by each center.
  60mL of blood is collected at baseline, 120mL annually, and 60mL at other events.
  Eligible individuals who are not seen in person for a clinic visit, who express interest in enrollment after initial contact, will be sent a copy of the IC document and a saliva collection kit by mail. Individuals in Cohort 5 may alternatively submit saliva or buccal swab samples without a clinic visit. Participants will return the signed consent and saliva sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Cohort 1: Individuals without history of PDAC meeting any of the following criteria:
  1. 2+ relatives with PDAC on same side of family where 2 affected are first degree related to each other and at least 1 affected is first degree related to subject; age 50+ or ≤10 years younger than earliest PDAC in family at time of diagnosis.
  2. 2 affected first degree relatives with PDAC; age 50+ or 10 years younger than earliest PDAC in family
  3. BRCA1, BRCA2, PALB2, ATM, MLH1, MSH2, MSH6, PMS2, EPCAM pathogenic or likely pathogenic variant AND 1 first or second degree relative with PDAC; age 50+ or 10 years younger than earliest PDAC in family
  4. Familial Atypical Moles and Malignant Melanoma (FAMMM) with pathogenic or likely pathogenic CDKN2A variant; age 40+
  5. Peutz-Jegher syndrome with STK11 pathogenic or likely pathogenic variant; age 35+
  6. Hereditary pancreatitis with PRSS1 pathogenic or likely pathogenic variant and history of pancreatitis; age 40+
- Cohort 2: Individuals without history of PDAC meeting any of the following criteria:
  1. ATM, BRCA1, BRCA2, or PALB2 pathogenic or likely pathogenic variant regardless of family history, age 50+
  2. 2+ relatives with PDAC on the same side of family, any degree of relation, not meeting other criteria above; age 50+ or 10 years younger than earliest PDAC in family
  3. 1 FDR with PDAC ≤ age 45; age up to 10 years younger than PDAC diagnosis in family member
- Cohort 3: Individual meeting criteria for Cohorts 1 or 2 EXCEPT age (i.e. too young to qualify for Cohorts 1 or 2)
- Cohort 4: Individuals without history of PDAC presenting for evaluation who do not meet any criteria for 1-3, 6, or the Cyst Cohort.
- Cohort 5: Individuals without history of PDAC who are not otherwise engaged in pancreas surveillance at a participating site may be invited to participate in the PRECEDE database and to donate a biosample (e.g. blood, saliva, and/or buccal swab) for discovery studies. This may include relatives of individuals in Cohorts 1-4,6, and the Cyst Cohort.
- Cyst Cohort: Individuals with a personal history of a pancreatic cystic neoplasm not meeting any criteria for Cohorts 1-3 or 6 (no known family history of PDAC, no known pathogenic germline variants linked to PDAC risk)
- Cohort 6a: Individuals diagnosed with PDAC or pancreatic high-grade dysplasia after enrollment in PRECEDE meeting any of the following criteria:
  1. Family history includes at least one first degree relative with PDAC, or 2 relatives with PDAC who are first degree related to each other
  2. Personal or family history of a pathogenic or likely pathogenic germline variant in ATM, BRCA1, BRCA2, CDKN2A, EPCAM, MLH1, MSH2, MSH6, PALB2,PMS2, PRSS1, STK11
- Cohort 6b: Individuals with a personal history of PDAC or pancreatic high-grade dysplasia meeting any of the following criteria:
  1. Family history includes at least one first degree relative with PDAC, or 2 relatives with PDAC who are first degree related to each other
  2. Personal or family history of a pathogenic or likely pathogenic germline variant in ATM, BRCA1, BRCA2, CDKN2A, EPCAM, MLH1, MSH2, MSH6, PALB2,PMS2, PRSS1, STK11
  3. Diagnosed ≤ age 45
- Cohort 6c: Individuals with newly diagnosed early stage (stage I or stage II) PDAC seen at a PRECEDE site that do not meet the criteria for 6a or 6b.
- Cohort 6d: Individuals with PDAC seen at a PRECEDE site that do not meet the criteria for 6a, 6b, or 6c.

SUMMARY:
The purpose of the Pancreatic Cancer Early Detection (PRECEDE) Consortium is to conduct research on multiple aspects of early detection and prevention of pancreatic ductal adenocarcinoma (PDAC) by establishing a multisite cohort of individuals with family history of PDAC and/or individuals carrying pathogenic/likely pathogenic germline variants (PGVs) in genes linked to PDAC risk for longitudinal follow up.

DETAILED DESCRIPTION:
The main objective of the PRECEDE Consortium is to build a shared resource to drive research in critical areas necessary for early detection and prevention of PDAC.

The PRECEDE Consortium is an observational prospective cohort study, with single or serial biosample collection (every 6-12 months) in defined high-risk groups.

A standardized procedure for collection and processing of human blood for the PRECEDE Consortium will be applied to all blood samples collected as part of the study. Barcoded samples will be stored at the clinical centers, using the specific labels for the PRECEDE study and corresponding data will be entered into the study database.

Clinical data and outcomes will be obtained from institutional databases or clinical records to correlate patient information with laboratory results from biospecimens obtained for research. Patients will be followed by their attending physician and receive the standard follow-up care after the procedure in which biospecimen was obtained. It is the intent that biospecimens will be made available to all consortium investigators.

ELIGIBILITY:
Inclusion Criteria:

Individuals from the following groups who present for clinical evaluation and assessment of PDAC risk at any of the participating sites can be offered participation in the PRECEDE database:

Cohort 1

Individuals without history of PDAC meeting any of the following criteria:

1. 2+ relatives with PDAC on same side of family where 2 affected are first degree related to each other and at least 1 affected is first degree related to subject; age 50+ or ≤10 years younger than earliest PDAC in family at time of diagnosis.
2. 2 affected first degree relatives with PDAC; age 50+ or 10 years younger than earliest PDAC in family
3. BRCA1, BRCA2, PALB2, ATM, MLH1, MSH2, MSH6, PMS2, EPCAM pathogenic or likely pathogenic variant AND 1 first or second degree relative with PDAC; age 50+ or 10 years younger than earliest PDAC in family
4. Familial Atypical Moles and Malignant Melanoma (FAMMM) with pathogenic or likely pathogenic CDKN2A variant; age 40+
5. Peutz-Jegher syndrome with STK11 pathogenic or likely pathogenic variant; age 35+
6. Hereditary pancreatitis with PRSS1 pathogenic or likely pathogenic variant and history of pancreatitis; age 40+

Cohort 2

Individuals without history of PDAC meeting any of the following criteria:

1. ATM, BRCA1, BRCA2, or PALB2 pathogenic or likely pathogenic variant regardless of family history, age 50+
2. 2+ relatives with PDAC on the same side of family, any degree of relation, not meeting other criteria above; age 50+ or 10 years younger than earliest PDAC in family
3. 1 first degree relative with PDAC ≤ age 45; age up to 10 years younger than PDAC diagnosis in family member

Cohort 3 Individual meeting criteria for Cohorts 1 or 2 EXCEPT age (i.e. too young to qualify for Cohorts 1 or 2)

Cohort 4 Individuals without history of PDAC presenting for evaluation who do not meet any criteria for 1-3, 6, or the Cyst Cohort.

Cohort 5 Individuals without history of PDAC who are not otherwise engaged in pancreas surveillance at a participating site may be invited to participate in the PRECEDE database and to donate a biosample (e.g. blood, saliva, and/or buccal swab) for discovery studies. This may include relatives of individuals in Cohorts 1-4,6, and the Cyst Cohort.

Cohort 6a

Individuals diagnosed with PDAC or pancreatic high-grade dysplasia after enrollment in PRECEDE meeting any of the following criteria:

1. Family history includes at least one first degree relative with PDAC, or 2 relatives with PDAC who are first degree related to each other
2. Personal or family history of a pathogenic or likely pathogenic germline variant in ATM, BRCA1, BRCA2, CDKN2A, EPCAM, MLH1, MSH2, MSH6, PALB2,PMS2, PRSS1, STK11

Cohort 6b

Individuals with a personal history of PDAC or pancreatic high-grade dysplasia meeting any of the following criteria:

1. Family history includes at least one first degree relative with PDAC, or 2 relatives with PDAC who are first degree related to each other
2. Personal or family history of a pathogenic or likely pathogenic germline variant in ATM, BRCA1, BRCA2, CDKN2A, EPCAM, MLH1, MSH2, MSH6, PALB2,PMS2, PRSS1, STK11
3. Diagnosed ≤ age 45

Cohort 6c Individuals with newly diagnosed early stage (stage I or stage II) PDAC seen at a PRECEDE site that do not meet the criteria for 6a or 6b.

Cohort 6d Individuals with PDAC seen at a PRECEDE site that do not meet the criteria for 6a, 6b, or 6c.

Cyst Cohort Individuals with a personal history of a pancreatic cystic neoplasm not meeting any criteria for Cohorts 1-3 or 6 (no known family history of PDAC, no known pathogenic germline variants linked to PDAC risk)

Exclusion Criteria:

* Individuals not meeting the criteria above.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will accrue subjects who present for risk assessment at one of the participating sites based on history of:
  * one or more family members with PDAC
  * a pathogenic or likely pathogenic germline variant in a gene linked to PDAC risk
  * personal history of PDAC with PGV in genes of research interest and/or part of a Familial Pancreatic Cancer kindred
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of PDAC | Through study completion, an average of 6 years
  Diagnosis of PDAC

CONTACTS AND LOCATIONS:
Overall Officials: Diane Simeone, MD, Study Chair — UC San Diego Moores Cancer Center
Locations (60):
- United States (45):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Honor Health Research Institute, Scottsdale, Arizona
  - Providence Health and Services, Burbank, California
  - City of Hope, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Health, Los Angeles, California
  - Hoag, Newport Beach, California
  - UC Irvine Health, Orange, California
  - UC Davis, Sacramento, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Illinois CancerCare, Bloomington, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Beaumont/Corewell Health, Royal Oak, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - White Plains Hospital, White Plains, New York
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (Upmc), Pittsburgh, Pennsylvania
  - University of Tennessee Graduate School of Medicine, Knoxville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Intermountain Health, St. George, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Epworth HealthCare, Richmond, Victoria, Australia
- Canada (3):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Semmelweis University, Institute of Pancreatic Diseases, Budapest, Hungary
- Landspitali University Hospital, Reykjavik, Iceland
- Sheba Medical Center, Ramat Gan, Israel
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy
- National Cancer Centre Singapore, Singapore, Singapore
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Arnau De Vilanova, Lleida
  - Ramón y Cajal University Hospital, Madrid
- Taiwan (2):
  - National Cheng Kung University Hospital (NCKUH), Tainan, Taiwan T.o.c.
  - National Taiwan University Hospital, Taipei
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zogopoulos G, Haimi I, Sanoba SA, Everett JN, Wang Y, Katona BW, Farrell JJ, Grossberg AJ, Paiella S, Klute KA, Bi Y, Wallace MB, Kwon RS, Stoffel EM, Wadlow RC, Sussman DA, Merchant NB, Permuth JB, Golan T, Raitses-Gurevich M, Lowy AM, Liau J, Jeter JM, Lindberg JM, Chung DC, Earl J, Brentnall TA, Schrader KA, Kaul V, Huang C, Chandarana H, Smerdon C, Graff JJ, Kastrinos F, Kupfer SS, Lucas AL, Sears RC, Brand RE, Parmigiani G, Simeone DM; PRECEDE Consortium. The Pancreatic Cancer Early Detection (PRECEDE) Study is a Global Effort to Drive Early Detection: Baseline Imaging Findings in High-Risk Individuals. J Natl Compr Canc Netw. 2024 Apr;22(3):158-166. doi: 10.6004/jnccn.2023.7097. PMID 38626807